CLINICAL TRIAL: NCT00031161
Title: Prevention of Dichloroacetate Toxicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: FD-R-2013-01; FD-R-002013-01
Record Dates: First submitted 2002-02-26; First posted 2002-02-27 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2002-01

CONDITIONS: Acidosis, Lactic; Chronic Disease
Keywords: Tyrosine; Diet; 2-(2-nitro-4-trifluoromethylbenzoyl)-1,3-cyclohexanedione; 4-Hydroxyphenylpyruvate Dioxygenase; Enzyme Inhibitors
MeSH Terms: conditions — Acidosis, Lactic; Chronic Disease | interventions — nitisinone; Dichloroacetic Acid

INTERVENTIONS:
Drug: Nitisinone (NTBC)
Drug: Dichloroacetate
Behavioral: Low-tyrosin diet

SUMMARY:
This is a study to determine the safety of dichloroacetate (DCA) with a low-tyrosine diet given with or without nitisinone (NTBC) in children with chronic lactic acidosis (CLA).

DETAILED DESCRIPTION:
DCA is being studied for the treatment of patients with CLA, which is a rare collection of mitochondrial metabolism errors causing cellular energy failure and early death. DCA causes reversible liver and peripheral nerve toxicity and it interrupts both tyrosine and heme metabolism. The inhibitory effect of DCA on mammalian tyrosine metabolism elicits biochemical changes similar to those observed in hereditary tyrosinemia type I (HT). However, some reports and studies indicate substantial reduction in the biochemical and clinical consequences of HT may occur when patients are treated concomitantly with a low-tyrosine diet (LTD) and the chemical NTBC, which inhibits an early step in tyrosine catabolism. Possibly, the same dietary and pharmacologic interventions may mitigate or prevent toxicity associated with chronic DCA exposure.

Patients visit the Center 5 times over a 1-year period, usually for 2 to 3 days per visit, for an extensive series of clinical and biochemical tests. Visit 1 is for baseline examinations and blood and urine chemistries and to educate the patient on an LTD. This visit lasts approximately 7 days to determine acceptable circulating tyrosine concentrations for LTD formula at discharge. Patients are provided with tubes to take to local laboratories every 2 weeks for blood work. Patients are readmitted in 1 month to determine adherence to diet and serum tyrosine levels. Patients who evidence dietary compliance, no adverse effects, and a willingness to continue are placed in 1 of 2 treatment arms: DCA plus an LTD plus placebo or DCA plus an LTD plus NTBC. Thereafter, patients return during Months 5, 9, and 13, which completes their 1-year treatment phase.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
Inclusion criteria:

* Biochemical or molecular genetic proof of a defect in mitochondrial enzyme of glucose metabolism or oxidative phosphorylation.
* Clinical history consistent with CLA (e.g., basal hyperlactatemia, stroke-like episodes, neuromuscular degeneration, and seizures).
* Ability to withstand an 8-hour fast (if 2 years old or younger) or a 12-hour fast without developing hypoglycemia (blood glucose greater than or equal to 50 mg/dL).

Exclusion criteria:

* Secondary lactic acidosis due to impaired oxygenation or circulation.
* Hyperlactatemia associated with proven biotinidase deficiency or with enzyme deficiencies of gluconeogenesis.
* Primary, defined organic acidurias other than lactic acidosis for which effective therapy is available (e.g., propionic aciduria).
* Primary disorders of amino acid metabolism.
* Primary disorders of fatty acid oxidation.
* Malabsorption syndromes associated with D-lactic acidosis.
* Renal insufficiency.
* Serum creatinine greater than 1.2 mg/g.
* Creatinine clearance less than or equal to 60 mL/min.
* Primary hepatic disease unrelated to chronic lactic acidosis.
* In patients with pyruvate dehydrogenase enzyme complex deficiency, an inability to maintain a diet greater than 50% calories from fat without biological and/or neurological deterioration.

Ages: 3 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2001-09; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States